CLINICAL TRIAL: NCT06206382
Title: Surgical Outcome of Borderline Resectable Pancreatic Cancer: Upfront Surgery Versus Neoadjuvant Chemotherapy (Single Center Experience)
Brief Title: Surgical Results of Resection of Locally Advanced Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Melad Boshra Yosef, Specialist, Assiut University
Other Study IDs: Borderline pancreatic cancer
Record Dates: First submitted 2024-01-02; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Upfront surgery for locally advanced pancreatic cancers
  Interventions: Procedure: Whipple operation
- Surgery after neoadjuvant chemotherapy for locally advanced pancreatic cancers
  Interventions: Procedure: Whipple operation

INTERVENTIONS:
Procedure: Whipple operation — Whipple operation is the surgery used for pancreatic head cancer in the form of pancreaticoduodenectomy then reconstruction

SUMMARY:
The aim is to compare the surgical outcomes between upfront surgery and surgery after neoadjuvant chemotherapy in terms of morbidity and mortality

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer death in the United States. While surgical resection remains the only curative option, more than 80% of patients present with unresectable disease. Unfortunately, even among those who undergo resection, the reported median survival is 15-23 mo, with a 5-year survival of approximately 20%. Disappointingly, over the past several decades, despite improvements in diagnostic imaging, surgical technique and chemotherapeutic options, only modest improvements in survival have been realized. Nevertheless, it remains clear that surgical resection is a prerequisite for achieving long-term survival and cure. The concept of borderline resectable pancreatic cancer has evolved from several clinical observations made over decades. It has been recognized for some time that the prognosis for patients undergoing surgical resection for pancreatic ductal adenocarcinoma (PDAC) is highly dependent on margin status, with total gross excision and histologically negative margins (R0 resection) being associated with the best outcomes. Survival for patients who undergo total gross excision but have histologically positive margins (R1 resection) have a reduced survival in most series

ELIGIBILITY:
Inclusion Criteria:

* Patients under surgical management for pancreatic cancer
* Patients whose radiological findings are compatible with resectability of the tumour including vascular encasement

Exclusion Criteria:

* Patients who are medically unfit for surgery
* Patients whose radioliogical findins suggestive of unresectability of the tumour including vascular abutment or infiltration more than 180 dergree

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of borderline respectable pancreatic cancer undergoing Whipple operation
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 years
  Patient death

SECONDARY OUTCOMES:
Morbidity | 6 months
  Surgical complications

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wang WL, Ye S, Yan S, Shen Y, Zhang M, Wu J, Zheng SS. Pancreaticoduodenectomy with portal vein/superior mesenteric vein resection for patients with pancreatic cancer with venous invasion. Hepatobiliary Pancreat Dis Int. 2015 Aug;14(4):429-35. doi: 10.1016/s1499-3872(15)60400-3. PMID 26256089
- [Background] Han S, Choi DW, Choi SH, Heo JS, Han IW, You YH. Long-term outcomes following en bloc resection for pancreatic ductal adenocarcinoma of the head with portomesenteric venous invasion. Asian J Surg. 2021 Jan;44(1):313-320. doi: 10.1016/j.asjsur.2020.07.021. Epub 2020 Sep 21. PMID 32972828
- [Background] Lapshyn H, Schulte T, Petruch N, Petrova E, Honselmann K, Deichmann S, Braun R, Kulemann B, Hoeppner J, Rades D, Keck T, Wellner UF, Bausch D, Bolm L. Postoperative Outcomes of Tangential versus Segmental Resection and End-to-end Reconstruction of the Superior Mesenterico-Portal Vein During Pancreatoduodenectomy for Pancreatic Adenocarcinoma: A Single-Center Experience. Anticancer Res. 2021 Oct;41(10):5123-5130. doi: 10.21873/anticanres.15329. PMID 34593463
- [Background] Yu XZ, Li J, Fu DL, Di Y, Yang F, Hao SJ, Jin C. Benefit from synchronous portal-superior mesenteric vein resection during pancreaticoduodenectomy for cancer: a meta-analysis. Eur J Surg Oncol. 2014 Apr;40(4):371-8. doi: 10.1016/j.ejso.2014.01.010. Epub 2014 Feb 7. PMID 24560302
- [Background] Tewari M. Significance of pathological positive superior mesenteric/portal venous invasion in pancreatic cancer. Hepatobiliary Pancreat Dis Int. 2016 Dec;15(6):572-578. doi: 10.1016/s1499-3872(16)60156-x. PMID 27919845